CLINICAL TRIAL: NCT02502773
Title: Fluid Loading in Abdominal Surgery: Saline Versus Hydroxyethyl Starch: A Double-blinded Multicenter Prospective Randomized Trial (FLASH Study)
Brief Title: Fluid Loading in Abdominal Surgery: Saline Versus Hydroxyethyl Starch (FLASH Study)
Acronym: FLASH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Agence Nationale de sécurité du Médicament (Other); Programme Hospitalier de Recherche Clinique (AOI N° 2013 _ Futier) (Unknown); Société Française Anesthesie-Réanimation (SFAR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0242; 2014-005575-84 (EudraCT Number)
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Morbidity; Postoperative Mortality
Keywords: Goal-directed therapy; Fluid loading; Abdominal surgery; Postoperative morbidity; Postoperative mortality; Individualized goal-directed fluid therapy; Elective or emergency abdominal surgery; General Anesthesia; Moderate-to-high risk surgical patients

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- crystalloid group (Experimental): The proposed Flash multicenter study will be conducted to assess if the use of HES or crystalloid solutions during an individualized GDT contribute to outcome differences in patients at moderate-to-high risk of postoperative complications after abdominal surgery
  Interventions: Drug: Hydroxethyl starch
- colloid group (Experimental): The proposed Flash multicenter study will be conducted to assess if the use of HES or crystalloid solutions during an individualized GDT contribute to outcome differences in patients at moderate-to-high risk of postoperative complications after abdominal surgery
  Interventions: Drug: Hydroxethyl starch

INTERVENTIONS:
Drug: Hydroxethyl starch

SUMMARY:
The primary purpose of the study is to evaluate whether the type of fluid (0.9% saline or 6% Hydroxyethyl starch 130/0.4) in the context of an individualized goal-directed fluid therapy is associated with a difference in morbidity and mortality within the first 14 days in patients at moderate-to-high risk of postoperative complications after abdominal surgery.

DETAILED DESCRIPTION:
Fluid administration is the mainstay treatment for suspected hypovolemia during surgery, but the effects of different crystalloid and colloid solutions on outcome remain poorly explored in surgical patients.

Two recent international multicenter studies (6S and CHEST studies) have shown that, compared to crystalloid solutions, the use of hydroxyethyl starch (HES) could be responsible for higher morbidity, especially renal failure, and mortality in ICU patients, thus leading to a recent restriction of their range of indications.

In contrast, in surgical patients, recent meta-analyses have concluded on the absence of difference in terms of mortality and postoperative renal failure between crystalloids and latest generation HES. Excessive fluid administration during surgery is associated with increased risk of postoperative morbidity, including renal dysfunction and mortality. It has been suggested that, compared with the volume-restoring effects of colloids, crystalloid use may require the administration of higher fluid volumes, which may contribute to poorer outcomes. In the surgical context, clinical trials and meta-analyses have shown that individualized goal-direct fluid administration can reduce postoperative morbidity. Although most GDT studies have used colloid solutions for fluid loading, the effects of the type of fluids are currently unknown and crystalloids are proposed for first-line therapy.

The proposed Flash multicenter study will be conducted to assess if the use of HES or crystalloid solutions during an individualized GDT contribute to outcome differences in patients at moderate-to-high risk of postoperative complications after abdominal surgery. As these fluids are widely used during surgery and because of current concerns about the risks related to the use of HES-based products in ICU patients, the trial will provide important data to clinicians involved in perioperative care.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who

* Undergo elective or emergency abdominal surgery under general anesthesia
* With an estimated surgical duration greater than or equal to 2 hours
* With moderate-to-high risk of postoperative complications defined by an AKI risk index≥ class 3, as defined by the presence of at least 4 of the following factors: age> 56 years, male gender, intraperitoneal surgery, active congestive heart failure, ascites, hypertension, emergency surgery, mild or moderate renal insufficiency, diabetes mellitus treated by oral or insulin therapy

Exclusion Criteria:

The following patients will not be evaluated for inclusion:

* Age <18 years
* Preoperative acute heart failure
* Preoperative acute coronary insufficiency
* Preoperative severe renal failure (defined by creatinine clearance <30 ml/min or requiring renal replacement therapy)
* Preoperative shock defined by the need for vasoactive amines
* History of allergy with the use of 6% Hydroxethyl starch 130/0.4
* Contraindication to the use of HES: sepsis, burnt patient, renal insufficiency or dialysis, cerebral hemorrhage, ICU patient , hypervolemia, lung edema, dehydration, severe hypernatremia or severe hyperchloremia, severe hepatic insufficiency, congestive heart failure, severe coagulopathy, organ transplant
* Patient's or relative's refusal to participate
* Parturient or breastfeeding woman
* Protected major (guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Renal dysfunction | during the first 14 postoperative days
  Renal dysfunction (defined by KDIGO stage 1 or higher)
Pulmonary complication | during the first 14 postoperative days
  Pulmonary complication (defined by the need for noninvasive or invasive ventilatory assistance for postoperative acute respiratory failure)
Cardiovascular complication | during the first 14 postoperative days
  Cardiovascular complication (defined by the development of acute heart failure)
Infectious complication | during the first 14 postoperative days
  Infectious complication (defined by the development of sepsis, severe sepsis or septic shock)
Surgical complication | during the first 14 postoperative days
  Surgical complication (defined as the need for surgical reoperation)

SECONDARY OUTCOMES:
Total fluid volume | during the surgical period and the first 24 postoperative hours
  Total fluid volume (0.9% saline and HES 130/0.4)
Volume of blood loss | during the surgical period and the first 24 postoperative hours
Renal complications : oliguria | within 14 days
  Postoperative complications
Cardiovascular complications | within 14 days
  Postoperative complications
Respiratory complications | within 14 days
  Postoperative complications
SIRS score | within 14 days
  Postoperative complications
Infectious complications | within 14 days
  Postoperative complications
Surgical complications | within 14 days
  Postoperative complications
Severity organ failure assessment score from postoperative | Day-1 to Day-7
Unexpected ICU admission (or readmission) following surgery | within 28 days
All-cause mortality | 28 days
All-cause mortality | 3 months
Serum lactate | from Day-1 to Day-7
C-reactive protein | from Day-1 to Day-7
Plasma chloride | from Day-1 to Day-7
number of units of packed red blood cells | during the surgical period and the first 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel FUTIER, Principal Investigator — University Hospital, Clermont-Ferrand; Jean-Etienne BAZIN, Principal Investigator — University Hospital, Clermont-Ferrand; Samir JABER, Principal Investigator — University Hospital, Montpellier; Julien POTTECHER, Principal Investigator — CHRU Strasbourg; Alexandre OUATTARA, Principal Investigator — University Hospital, Bordeaux; Thomas LESCOT, Principal Investigator — Hôpital Saint-Antoine (APHP); Hélène BELOEIL, Principal Investigator — CHU Rennes; Gilles LEBUFFE, Principal Investigator — CHRU LILLE; Philippe CUVILLON, Principal Investigator — CHU Nîmes; Julien BUREY, Principal Investigator — Hôpital Tenon (APHP); Willy-Serge MFAM, Principal Investigator — CH ORLEANS; Vincent PIRIOU, Principal Investigator — Hospices Civils de Lyon; Marc LEONE, Principal Investigator — AP-HM; Sébastien BERTRAN, Principal Investigator — CHU Nîmes; Marion FAUCHER, Principal Investigator — Institut Paoli-Calmettes; Catherine PAUGAM-BURTZ, Principal Investigator — Hôpital Beaujon; Lionel VELLY, Principal Investigator — AP-HM; Olivier HUET, Principal Investigator — CHU Brest; Sigismond LASOCKI, Principal Investigator — University Hospital, Angers; Pierre SAINT-LEGER, Principal Investigator — CH VALENCIENNES
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Futier E, Garot M, Godet T, Biais M, Verzilli D, Ouattara A, Huet O, Lescot T, Lebuffe G, Dewitte A, Cadic A, Restoux A, Asehnoune K, Paugam-Burtz C, Cuvillon P, Faucher M, Vaisse C, El Amine Y, Beloeil H, Leone M, Noll E, Piriou V, Lasocki S, Bazin JE, Pereira B, Jaber S; FLASH Trial Group; Lasocki S, Huet O, Cadic A, Jacob C, Paugam-Burtz C, Restoux A, Ouattara A, Feitita I, Deloge E, Defaye M, Joannes-Boyau O, Carles P, Napolitano G, Monziols S, Futier E, Vignaud M, Paul S, Gahbiche K, Fayon J, Laroche E, Bazin JE, Brandely A, Le Moal C, Lebuffe G, Garot M, Piriou V, Jaber S, Chanques G, Verzilli D, De Jong A, Millot A, Castagnoli A, Leone M, Pastene B, Castelli C, Medam S, Velly L, Vaisse C, Faucher M, Asehnoune K, Samba E, Roquilly A, Le Penndu M, Cuvillon P, Yves Lefrant J, Wira O, Dubout E, Mfam WS, Lescot T, Begneu E, Burey J, Cirilovic T, Beloeil H, Allo G, Pottecher J, Lebas B, Venot C, Rameau JP, Dimache F, Leger PS, El Amine Y. Effect of Hydroxyethyl Starch vs Saline for Volume Replacement Therapy on Death or Postoperative Complications Among High-Risk Patients Undergoing Major Abdominal Surgery: The FLASH Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):225-236. doi: 10.1001/jama.2019.20833. PMID 31961418
- [Derived] Futier E, Biais M, Godet T, Bernard L, Rolhion C, Bourdier J, Morand D, Pereira B, Jaber S; FLASH trial management committee. Fluid loading in abdominal surgery - saline versus hydroxyethyl starch (FLASH Trial): study protocol for a randomized controlled trial. Trials. 2015 Dec 21;16:582. doi: 10.1186/s13063-015-1085-3. PMID 26690683